CLINICAL TRIAL: NCT06705504
Title: Real-world Effectiveness and Safety in HR+/HER2- Advanced or Metastatic BC Patients Treated With Ribociclib or Alpelisib: A European Non-interventional Retrospective Study (REASSURE)
Brief Title: A Real-world Study of Effectiveness and Safety in HR+/HER2- Breast Cancer Patients Treated With Ribociclib or Alpelisib
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CLEE011A3002
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hormone Receptor Positive HER-2 Negative Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Institut de Cancérologie de l'Ouest (ICO) Cohort: Patients with HR+/HER2- advanced or metastatic BC who were registered in IQVIA's oncology evidence network (OEN), ICO, and initiated treatment with ribociclib or alpelisib.
- L'Institut Curie (Curie) Cohort: Patients with HR+/HER2- advanced or metastatic BC who were registered in IQVIA's OEN, Curie, and initiated treatment with ribociclib or alpelisib.
- Instituto Português de Oncologia do Porto (IPO-Porto) Cohort: Patients with HR+/HER2- advanced or metastatic BC who were registered in IQVIA's OEN, IPO-Porto, and initiated treatment with ribociclib or alpelisib.
- Czech Republic Cohort: Patients with HR+/HER2- advanced or metastatic BC who were registered in Czech Republic local sites or clinics proposed by Novartis affiliates and initiated treatment with ribociclib or alpelisib.

SUMMARY:
This study was a multinational and multicenter cohort study of patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative (HR+/HER2-) advanced or metastatic breast cancer (aBC/mBC) treated with ribociclib or alpelisib between the period of 01 January 2018 and 30 September 2021. Patients who were receiving active treatment for malignancies other than BC or participating in a clinical trial were excluded. This study was conducted retrospectively with secondary use of data.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of locally advanced/metastatic not amenable to surgery HR+/HER2- BC (progressed following prior therapy or de novo) for whom the treating physician took the decision to initiate treatment with ribociclib or alpelisib.
* Patients with at least one prescription for ribociclib or alpelisib during the index period (01 January 2018 to 30 September 2021).

Exclusion criteria:

* Patients who were participating in any interventional clinical trial that included investigational or marketed products at the time of index (ribociclib, alpelisib, and other); patients who were participating in other investigator-initiated research or non-interventional study (NIS) could be included as long as their standard of care was not altered by the study.
* Patients on active treatment for malignancies other than HR+/HER2- aBC/mBC at the time of index.
* IPO-Porto cohort only:

  * Patients who had participated or were participating in any interventional clinical trial that included investigational or marketed products at the time of index (ribociclib, alpelisib, and others).
  * Patients who underwent part of the treatment for locally advanced/metastatic not amenable to surgery HR+/HER2- BC outside the center.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Real-world Progression-free Survival (rwPFS) | Up to 51 months
  rwPFS was defined as the time from the index date to the date of the first documented progression or death due to any cause. If a patient did not have an event, rwPFS was censored at the date of the last adequate tumor assessment. The index date was defined as the date of the first treatment with ribociclib or alpelisib.

SECONDARY OUTCOMES:
Age | Baseline
Number of Patients by Age Group | Baseline
  Age groups:
  * Younger than 65 years
  * 65 years or older
Gender | Baseline
Number of Patients Categorized by Year of Index Date | Baseline
  The index date was defined as the date of the first treatment with ribociclib or alpelisib.
Number of Patients With a History of Breast Cancer | Baseline
Number of Patients by Comorbidity | Baseline
  Comorbidities included:
  * Diabetes mellitus
  * Cardiovascular disease
  * Cerebrovascular disease
  * Chronic obstructive pulmonary disease (COPD)
  * Dementia
  * Depression
  * Heart Failure
  * Hypertension
  * Hypothyroidism
  * Ischemic heart disease
  * Liver disease
  * Myocardial infarction
  * Osteoporosis
  * Peripheral vascular disease
  * Renal Disease
  * Rheumatological disease
  * Ulcer disease
  * Other
Body Mass Index (BMI) | Baseline
Number of Patients per BMI Category | Baseline
  BMI Categories:
  * Underweight: below 18.5 kilograms per meter squared (kg/m^2)
  * Healthy/normal weight: 18.5 to 24.9 kg/m^2
  * Pre-obesity: 25 to 29.9 kg/m^2
  * Obesity: 30 kg/m^2 and higher
Number of Patients by Menopausal Status | Baseline
  Menopausal status:
  * Pre- or peri-menopausal
  * Post-menopausal
Number of patients per Charlson Comorbidity Index (CCI) Score Category | Baseline
  CCI predicts the ten-year mortality for a patient who may have a range of comorbid conditions. Comorbidity was assessed using the CCI, categorized as low (0-1) and high (≥2).
Number of Patients Categorized by Duration of Disease Recurrence | Baseline
  Disease recurrence categories:
  * 12 months or less
  * More than 12 months
Number of Patients by Smoking Status | Baseline
  Smoking status:
  * Current smoker
  * Former smoker
  * Never smoked
Number of Patients Categorized by Primary Tumor Type | Baseline
  Tumor types:
  * Invasive ductal
  * Lobular carcinoma
  * Other
Number of Patients Categorized by Disease Site | Baseline
  Disease site categories:
  * Non-visceral
  * Visceral
  * Multiple
Number of Patients With Primary Metastatic Disease | Baseline
Number of Patients Categorized by Number of Metastatic Sites | Baseline
  Categories for number of metastatic sites: 0, 1, 2, 3, 4 or more.
Number of Patients Categorized by Type of Metastases | Baseline
  Metastases:
  * Local/breast metastases
  * Bone metastases
  * Lung metastases
  * Liver metastases
  * Central nervous system metastases
  * Lymph node metastases
  * Other metastases
Number of Patients Categorized by Time From Diagnosis to Metastasis | Baseline
  Categories:
  * 24 months or less
  * More than 24 months
  * Metastatic BC at diagnosis
Number of Patients With Asymptomatic Disease | Baseline
Number of Patients Categorized by Tumor Grade | Baseline
  Tumor Grades:
  * Grade 1
  * Grade 2
  * Grade 3
Number of Patients Categorized by Stage of Cancer | Baseline
  Cancer Stages: I, IIA, IIB, IIIA, IIIB, IIIC, and IV.
Number of Patients by Eastern Cooperative Oncology Group (ECOG) Performance Score | Baseline
  ECOG performance score describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Scores ranged from a lower value of 0 (fully active, able to carry out all pre-disease performance without restriction) up to 4 (completely disabled; cannot carry out any selfcare; totally confined to bed or chair).
Number of Patients Categorized by Previous Types of Treatment | Baseline
  Treatment categories:
  * Chemotherapy
  * Surgery
  * Radiotherapy
  * Adjuvant endocrine therapy
  * Everolimus treatment
Number of Patients Categorized by the Number of Prior Lines of Endocrine Therapy (ET) | Baseline
  Categories for number of lines of ET: 0, 1, 2, and 3 or more.
Number of Patients Resistant to ET | Baseline
Number of Patients Sensitive to Hormonal Therapy | Baseline
Number of Patients Categorized by Line of Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) Treatment Received | Baseline
  CDK4/6i lines of treatment:
  * Adjuvant
  * 1st metastatic line
  * 2nd metastatic line
  * 3rd metastatic line or later
Number of Patients Categorized by the Number of Previous Lines of Treatment | Baseline
  Categories for number of lines of treatment: 0, 1, 2, and 3 or more.
Baseline Neutrophil-to-lymphocyte Ratio (NLr) | Baseline
Baseline Platelet-to-lymphocyte Ratio (PLr) | Baseline
Baseline Lymphocytes-to-monocytes Ratio (LMr) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States